CLINICAL TRIAL: NCT03263455
Title: The Effects of Kinesis-Taping Application on Cognitive Deficit and Motor Ability in Stroke Patients With Visuospatial Neglect: a Randomized Controlled Study
Brief Title: Kinesio-Taping in Stroke Patients With Visuospatial Neglect
Acronym: k-neglect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Full Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KN2017
Record Dates: First submitted 2017-08-14; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Stroke; Motor Disorder
Keywords: neglect,; stroke,; rehabilitation,; range of motion
MeSH Terms: conditions — Stroke; Motor Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping group (Experimental): The tape in the KT group was applied with paper-off tension, which means applying the tape directly to the skin as it comes off the paper backing (approximately with 15% to 25% of available tension).
  Interventions: Other: Kinesio taping group
- Sham Taping group (Sham Comparator): Patients in the ST group, smaller "I-strips" of KinesioTape were used and they were applied, with no tension and without stretching the muscles, perpendicularly to the muscle belly (starting from the middle and progressing to each side) over the same dystonic muscles as in the Kinesio Taping group
  Interventions: Other: Sham Taping

INTERVENTIONS:
Other: Kinesio taping group — The tape in the KT group will be applied with paper-off tension, which means applying the tape directly to the skin as it comes off the paper backing (approximately with 15% to 25% of available tension). KinesioTape will be applied over the SCM dystonic muscle by means of 2 "I-strips": the first strip will be placed on the medial (sternal) head and the second will be applied on the lateral (clavicular) head of the SCM muscle. KinesioTape was applied from the mastoid bone to the clavicle (rostrocaudal direction) with the SCM placed in a position of maximum stretching.
  Arms: Kinesio Taping group
Other: Sham Taping — Patients in the ST group, smaller "I-strips" of KinesioTape will be used and they will be applied, with no tension and without stretching the muscles, perpendicularly to the muscle belly (starting from the middle and progressing to each side) over the same dystonic muscles as in the experimental group. Although the specific therapeutic elements of KinesioTaping (ie, longitudinal stretch, start and ending point tape application) will be removed
  Arms: Sham Taping group

SUMMARY:
Stroke is the second leading cause of death worldwide and the third most common cause of disability. The effects of stroke are variable and may include impairments in motor and sensory systems, emotion and neuropsychological deficits such as a disorder of spatial awareness known as unilateral spatial neglect (USN). Approaches to ameliorate USN could be categorized in interventions as involving either bottom-up or top-down processing. The specific mechanisms underlying these effects on a number of manifestations of the USN syndrome may include the restoration of defective representations of the side of space contralateral to the lesion (contralesional), and of the ability to orient spatial attention contralesionally, through complex patterns of activation of both the damaged right hemisphere, and the contralateral left hemisphere, with differences related to the specific stimulation delivered to the patient. In recent years, increasing cutaneous stimuli through neuromuscular kinesiotaping has been proposed to enhance somatosensory inputs (24) and such as method could have positive effects on USN. The aim of the present study was to assess the effect of KTM applied on the sternocleidomastoid muscle controlateral side of the lesions in improving USN deficits in individuals with stroke patient in sub-acute phase. The hypothesis is that the KTM application could improved cognitive tests for assessing USN, motor deficits and kinesthetic neck sensibility.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by stroke from cerebral ischemia or hemorrhage that occurred ⩽ 30 days before;
* presence of visuospatial neglect (Star Cancellation Test' score < 50)
* able to actively rotate the head toward left side in closed eyes condition.

Exclusion Criteria:

* the presence of dementia (Mini-Mental State Examination correct score lower than 23,80)
* severe deficit of comprehension
* psychiatric disorders
* hemianopsia patients (diagnosed with perimetry) patients or their family members did not consent to this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2017-11-30 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
The Stars Cancellation Test change in number of stars deleted | Baseline time 0 and up to 4 weeks

SECONDARY OUTCOMES:
Number of letter delete during the Letter Cancellation Test | Baseline time 0 and up to 4 weeks
Number of Error assessed during the Cervical Joint Position Error Test | Baseline time 0 and up to 4 weeks
Degree of Active Range of Motion (AROM) during left rotation | Baseline time 0 and up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Smania, MD, Principal Investigator — Neuromotor and Cognitive Rehabilitation Center Department for Neurosciences, Biomedicine and Movement Sciences University of Verona, Verona, Italy P.zza L.A. Scuro, 10 37134 Verona, Italia; Alessandro Picelli, MD, Study Director — Neuromotor and Cognitive Rehabilitation Center Department for Neurosciences, Biomedicine and Movement Sciences University of Verona, Verona, Italy P.zza L.A. Scuro, 10 37134 Verona, Italia
Locations (2):
- Italy (2):
  - Azienta Ospedaliera, SSO Rehabilitation Unit, Verona, Verona, Italy, Verona
  - Azienta Ospedaliera, SSO Rehabilitation Unit, Verona, Verona

IPD SHARING:
Plan to Share IPD: No